CLINICAL TRIAL: NCT06407804
Title: Effects of Thrower's Ten and Routine Physical Therapy on Pain, Range of Motion and Functional Disability in Patients With Shoulder Impingement Syndrome
Brief Title: Effects of Thrower's Ten and Routine Physical Therapy in Patients With Shoulder Impingement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01110
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrower's Ten Exercise Program (Experimental): 1. D2 PNF flexion
  2. D2 PNF extension
  3. Internal rotation
  4. External rotation
  5. Push ups
  6. Press ups
  Interventions: Other: Thrower's Ten Exercise Program
- Routine physical therapy (Sham Comparator): 1. Unilateral bench press
  2. Bi lateral shoulder retraction
  3. Extension in prone position
  4. Neck retraction. Then isometrics will be performed which includes
  1. Isometric shoulder internal and external rotation 2. Side lying shoulder external rotation 3. Scapular scaption exercise
  Interventions: Other: Routine physical therapy.

INTERVENTIONS:
Other: Thrower's Ten Exercise Program — No Of Sessions Per Week: 3 Per Weeks for 6 weeks (50 Min per Session) No of repetitions; 2 sets for 10 repetitions with 1 minute rest between sets.
  Other Names: Routine physical therapy
  Arms: Thrower's Ten Exercise Program
Other: Routine physical therapy. — In this, the exercises will be performed in 2 sets and 10 repetitions with 5-10s hold and 30s to 1min rest between repetitions.
  No Of Sessions Per Week: 3 Per Weeks for 6 weeks (50 Min Per Session)
  Arms: Routine physical therapy

SUMMARY:
To compare the effects of thrower's ten and routine physical therapy on pain, range of motion and functional disability in patients with shoulder impingement syndrome

DETAILED DESCRIPTION:
Shoulder impingement is a common cause of shoulder pain. It's also known as impingement syndrome or swimmer's shoulder, since it's common in swimmers. It occurs when there is impingement of tendons or bursa in the shoulder from bones of the shoulder. A randomized clinical trial will be conducted at Ibne Sina Hospital,Multan . Non probability convenience sampling technique will be applied on 46 patients who will be allocated through computerized randomization into group A & group B to collect data. Group A will be given Throwers ten Program and group B will be given routine physical therapy along with baselines. The study will be completed within the time duration of nine months. Primary Outcome measures of the research will be pain, range of motion,function and disability . Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-35 years
* Male and female
* Shoulder or neck pain within the prior 6month
* 3 positive tests out of 5: Positive Neer's test, positive Hawkins test, positive Jobe's test, painful arc, and pain on resisted external rotation of the arm.

Exclusion Criteria:

* History of surgery of the affected shoulder
* Fractures in around the shoulder
* Neurological disorders leading to altered muscle activity
* Systemic arthritic conditions (RA, Osteoporosis)
* Disorders of the cervical spine

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  The Numeric Pain Rating Scale (NPRS) is used to assess pain. On an 11-point Numeric scale, 0 represents the least amount of pain (no pain) and 10 Represents the most amount of pain (worst pain)
Range of Motion | 6 weeks
  It is frequently employed as a benchmark technique for the assessment of Range of Motion (ROM) as the main component of all joint motions. The range of mobility of a joint is measured using a device known as a goniometer. Goniometry is the art and science of measuring the joint ranges in every plane of the joint. Short arm and long arm versions of the universal goniometer are available. Goniometric measurements are highly reliable provided measurements are conducted by the same therapist. Shoulder Abduction, Flexion and External rotation range will be taken by a Universal Goniometer.
Shoulder pain and disability index (SPADI) | 6 weeks
  The SPADI (Shoulder Pain and impairment Index) was created to assess current shoulder pain and impairment in an outpatient environment. The SPADI consists of 13 items that assess two domains: a 5-item subscale for pain and an 8-item subscale for disability. The SPADI has since been used in both primary care on mixed diagnosis and surgical patient populations including rotator cuff disease, osteoarthritis, and rheumatoid arthritis, adhesive capsulitis ,joint replacement surgery , and in a large population-based study of shoulder symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Johar Pain Relief Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No